CLINICAL TRIAL: NCT01272518
Title: Assessment of Cardiac Autonomic Behavior in Patients With Mood Disorders With a Focus on the Chaos Theory
Brief Title: Assessment of Cardiac Autonomic Behavior in Patients With Mood Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sao Jose do Rio Preto Medical School (Other)
Responsible Party: Principal Investigator, Guilherme Luiz, Guilherme Luiz Lopes Wazen, Sao Jose do Rio Preto Medical School
Other Study IDs: 459/2010; sao jose RPU (Registry Identifier: 459/2010)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Mood Disorder; Mania; Depression
Keywords: chaos theory heart rate variability mania bipolar disorder
MeSH Terms: conditions — Mood Disorders; Mania; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to characterize the behavior of cardiac patients with Mood Disorders and its clinical course, interpreting the results from a theoretical framework of Chaos Theory and Complexity Theory and Systems as well.

DETAILED DESCRIPTION:
Mood disorders are strongly associated with changes in cardiovascular function and alterations in Hear Rate Variability (HRV). Fluctuation in heart rate occurs over a wide frequency and demonstrates a broad, irregular variability that suggests that the mechanisms involved in cardiovascular regulation interact in a nonlinear manner. Over the past decade, there has been an increasing emphasis on applying nonlinear methods of analysis to characterize cardiac function, but the studies on the pathophysiology of mood disorders in general still remain under a linear and reductionist perspective. The scarcity of both Brazilian and international studies on the autonomic behavior in mood disorders in general and not only in Major Depressive Disorder, as well as the use of a non-linear reading of the results of this study makes an additional tool of analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Bipolar Disorder (BD) or Major Depressive Disorder(MDD)

Exclusion Criteria:

* Another with criteria for Axis I or II disorders aside from the primary diagnosis of BD or MDD.
* Past history of stroke, heart attack, or cardiac disease.
* Drug abuse or dependence in the past six months.
* Diabetes.
* In use of Tricyclic Antidepressants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely hospitalized patient and in ambulatorial attendance with Bipolar Disorder or Major Depressive Disorder.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression(HAM-D-17)-17 ; Montgomery & Asberg Rating Scale for Depression(MADRS); Escala de Avaliação de Mania de Bech-Rafaelsen (EAM-BR); Mini International Neuropsychiatric Interview (MINI. | 3 months (period between the first and the second assessments)
  Both scales for depression and mania will be compared with the linear and nonlinear results from the heart rate variability in the period of 3 months.

SECONDARY OUTCOMES:
Polar RS800CX hear-rate monitor; Kubios HRV version 2.0 software; Visual Recurrence Analysis software. | 3 months (period between the first and the second assessments)
  The heart rate variability will be obtained from 20-min R to R wave (RR) interval data using the Polar. The data will be estimated by analysis from both softwares.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme L Wazen, Principal Investigator — São José do Rio Preto Faculty of Medicine (FAMERP) / Departament of Psychiatry - FAMERP / NUTECC (Nucleo Transdisciplinar para Estudo do Caos e da Complexidade); Moacir F Godoy, Professor, Study Director — São José do Rio Preto Faculty of Medicine (FAMERP) /Cardiology and Cardiovascular Surgery Department -FAMERP/ NUTECC (Nucleo Transdisciplinar para Estudo do Caos e da Complexidade)
Locations (1):
- São José do Rio Preto Faculty of Medicine, São José do Rio Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Gregorio ML, Wazen GLL, Kemp AH, Milan-Mattos JC, Porta A, Catai AM, de Godoy MF. Non-linear analysis of the heart rate variability in characterization of manic and euthymic phases of bipolar disorder. J Affect Disord. 2020 Oct 1;275:136-144. doi: 10.1016/j.jad.2020.07.012. Epub 2020 Jul 10. PMID 32658816